CLINICAL TRIAL: NCT02182466
Title: Documentation of Colon Capsule Endoscopies in a National Observational Study [Dokumentation Von Kolonkapsel-Endoskopien im Rahmen Einer Bundesweiten Studie]
Brief Title: German Colon Capsule Registry
Acronym: DEKOR
Status: Terminated | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Jorg Albert, [Dokumentation von Kolonkapsel-Endoskopien im Rahmen einer bundesweiten Studie], Johann Wolfgang Goethe University Hospital
Other Study IDs: 265/13; DRKS-ID: DRKS00006283 (Other: German Clinical Trials Registry)
Record Dates: First submitted 2014-06-27; First posted 2014-07-08 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Colon Cancer; Colon Polyp; Diarrhea; Inflammatory Bowel System; Ulcerative Colitis
Keywords: Colon capsule endoscopy; Colonoscopy; Screening colonoscopy
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps; Diarrhea; Colitis, Ulcerative | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colonic endoscopy indicated
  Interventions: Device: Colon capsule endoscopy

INTERVENTIONS:
Device: Colon capsule endoscopy

SUMMARY:
Aim of the registry is to evaluate all colon capsule endoscopies performed in Germany. This is to investigate safety, quality assurance and quality control of colon capsule endoscopy.

DETAILED DESCRIPTION:
Colon capsule endoscopy (CCE, Pill Cam Colon 2, (Given Imaging Ltd, Yoqneam, Israel and Given Imaging EMEA, Hamburg, Germany) provides direct visualization of the colon mucosa, enabling the investigator to diagnose colonic disease. CCE is a complementary means to flexible ileo-colonoscopy andt safety, quality assurance and quality control of CCE is not well understood. There are about 15 000 investigations performed worldwide until now, but systematic data on performance in a community based setting are lacking.

This study aims to investigate safety, quality assurance and quality control of colon capsule endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Indication for colon capsule endoscopy
* Age of 18 years or older
* Consent of the patient

Exclusion Criteria:

* Intestinal obstruction
* Dyphagia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication for endoscopic investigation of the colon
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-06; Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Establishing a diagnosis from colon capsule endoscopy | At presentation of the patient until dismissal from medical care, an expected average of 2 weeks after performance of the investigation
  Participants will be followed for the time of presentation at the outpatient clinic or for the duration of hospital stay, an expected average of 2 weeks after performance of the investigation

SECONDARY OUTCOMES:
Technical success of colon capsule endoscopy | At presentation of the patient for performing colon capsule endoscopy until end of colon capsule endoscopy, an average of 24 hours
  Technical success is evaluated during the investigation and immediately after to identifal correct technical function of the capsule endoscope including technical performance of the system, battery life of the capsule, passage of colon capsule, review of the capsule video, and documentation
Complications of colon capsule endoscopy, i.e. number of participants with Adverse Events and characterization of Adverse Events | At presentation of the patient until dismissal from medical care, an expected average of 2 weeks after performance of the investigation
  Participants will be followed for the time of presentation at the outpatient clinic or for the duration of hospital stay. Thereby, participants with adverse events attributable to colon capsule endoscopy are assessed and AE characterized.
Cleansing level of colon capsule endoscopy | At presentation of the patient until dismissal from medical care, an expected average of 2 weeks after performance of the investigation
  Cleansing level of the colon is assessed and qualified as adequate or as not adequate.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg G Albert, MD, Principal Investigator — Frankfurt University Hospital Department of Internal Medicine I Theodor-Stern-Kai 7 D-60590 Frankfurt/Main Germany
Locations (1):
- Frankfurt University Hospital, Frankfurt am Main, Hesse, Germany